CLINICAL TRIAL: NCT00525460
Title: A Pilot Study of Young Women Diagnosed With Early Stage Ovarian Cancer: A Focus on Fertility Issues and Sexual Function
Brief Title: Young Women Diagnosed With Early Stage Ovarian Cancer: A Focus on Fertility Issues and Sexual Function
Status: Completed | Type: Observational
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Susana M. Campos, MD, Medical Oncologist, Dana-Farber Cancer Institute
Other Study IDs: 05-382
Record Dates: First submitted 2007-09-04; First posted 2007-09-05 (Estimated); Last update posted 2018-07-27 (Actual); Status verified 2018-07

CONDITIONS: Ovarian Cancer
Keywords: fertility; stage I ovarian cancer; stage II ovarian cancer; fertility sparing
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Fertility-Sparing Survey — A questionnaire completed either in the clinic or at home

SUMMARY:
The purpose of this study is to ask youn women diagnosed with ovarian cancer who have undergone surgery that will allow them to have children in the future, on issues such as: education about their options to keep their ability to have children, after-chemotherapy treatment decision making, and reproductive history. The second purpose is to determine the effect of an early diagnosis of ovarian cancer on the sexual functioning of women.

DETAILED DESCRIPTION:
* Participants will be asked to complete a questionnaire either in the clinic or at home and return it to the research staff by mail or in person.
* The study will involve being asked questions about the following: Fertility history; sexual history after being diagnosed with cancer; decision to have surgery that will allow them to have children; education they may or may not have received about the surgery that saved their ability to have children.
* Answers to all questions will be kept confidential and participants will be identified by a number only.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with stage I or II invasive ovarian cancer, that underwent fertility sparing surgery
* Women who were premenopausal prior to diagnosis
* 40 years of age or younger at the time of ovarian cancer diagnosis
* Completed therapy for early stage cancer
* No evidence of recurrence
* No history fo known infertility prior to diagnosis
* No other significant medical conditions that would affect fertility

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women 40 years of age or younger when diagnosed with ovarian cancer who chose to have surgery that allowed them to keep their reproductive organs
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2006-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To survey young women diagnosed with ovarian cancer who have undergone fertility sparing surgery on issues such as fertility counseling, post treatment decision making and reproductive history. | 36 months

SECONDARY OUTCOMES:
To determine the effect of an early diagnosis of ovarian cancer on the sexual functioning of women. | 36 months
To determine the feasibility of the Fertility-Sparing Survey included in this study. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Susana Campos, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts